CLINICAL TRIAL: NCT05926401
Title: Atrial Fibrillation Prior and Post Elective Cardioversion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 543834
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Planned elective cardioversion for atrial fibrillation
  Interventions: Other: ECG monitoring prior and after cardioversion

INTERVENTIONS:
Other: ECG monitoring prior and after cardioversion — Continuous ECG monitoring at home 3-5 days prior to and 5-7 days after planned cardioversion

SUMMARY:
Cardioversion from atrial fibrillation (AF) to sinus rhythm (SR) is performed primarily to improve patient symptoms. However, due to the intermittent nature of AF, patients may have converted to SR prior to elective cardioversion and the recurrence rate of AF after cardioversion can be high. The aims of this study are to assess the rate of spontaneously conversion to SR in patients with AF scheduled for elective cardioversion, as well as the rate of early recurrence of AF after elective cardioversion.

ELIGIBILITY:
Inclusion Criteria:

* Planned elective cardioversion of AF
* Informed written consent for participation

Exclusion Criteria:

* Lack of ability to cooperate
* Pacemaker/CRT device
* No smart phone

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients satisfying the inclusion criteria will be recruited after informed written consent for study participation.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of spontaneously conversion to SR in patients with AF scheduled for elective cardioversion | 10 days pre/post cardioversion
The rate of early recurrence (<5 days) of AF after elective cardioversion | up to 5 days pre/post cardioversion

CONTACTS AND LOCATIONS:
Overall Officials: Sigrun Halvorsen, PhD, Study Chair — Oslo university hospital /University of Oslo
Locations (1):
- Sorlandet Hospital, Arendal, Norway

IPD SHARING:
Plan to Share IPD: No